CLINICAL TRIAL: NCT00322920
Title: A Phase I Study of Weekly Topotecan With Cisplatin for the Management of Advanced Stage or Recurrent Carcinoma of the Cervix
Brief Title: Efficacy Study of Weekly Topotecan With Cisplatin in Advanced Stage or Recurrent Cervical Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low accrual
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: GlaxoSmithKline (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 104799
Record Dates: First submitted 2006-05-05; First posted 2006-05-08 (Estimated); Last update posted 2008-02-15 (Estimated); Status verified 2008-02

CONDITIONS: Cervix Cancer
Keywords: cervical cancer; topotecan; Stage IVB cervical cancer; Persistent or recurrent cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Topotecan; Cisplatin

INTERVENTIONS:
Drug: Topotecan
Drug: Cisplatin

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose (MTD) of topotecan when given weekly with cisplatin in patients with persistent, recurrent, or advanced stage cervical cancer. Secondary purposes are to describe the toxicity profile in patients with persistent, recurrent, or advanced stage cervical cancer treated with the combination of topotecan when given weekly with cisplatin and to determine the response rate and time to progression in patients with persistent, recurrent, or advanced stage cervical cancer treated with the combination of topotecan when given weekly with cisplatin.

DETAILED DESCRIPTION:
Patients diagnosed with recurrent cervical cancer generally have limited options for cure. Occasionally, radiation therapy may be utilized in localized recurrent disease with curative intent; however, most patients are not candidates for curative therapy secondary to disseminated disease, and thus are frequently treated with palliative chemotherapy. Initial experiences with chemotherapy in this clinical setting demonstrated cisplatin to be an active agent. Subsequent trials using combinations of cisplatin and ifosfamide or paclitaxel demonstrated higher response rates compared to cisplatin alone but did not demonstrate an improvement in overall survival. Topotecan is a topoisomerase I inhibitor that has been used in the management of cervical and ovarian cancer. Several phase II studies have demonstrated topotecan to be an active agent in cervical cancer. In an effort to ameliorate toxicity noted with 3-5 day dosing regimens of topotecan, investigators have evaluated weekly dosing of topotecan. Thus far, the toxicity of weekly topotecan dosing in cervical cancer has not been evaluated. In this study, topotecan will be given weekly at escalating dose levels starting at 2.0 mb/m2 with standard cisplatin at 50 mg/m2 every 21 days. This study will help to determine acceptable dosing for the combination of weekly topotecan and cisplatin in patients with persistent, recurrent, or advanced stage cervical cancer which can then be utilized in a cohort of patients with cervical cancer in a phase II study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have persistent, recurrent, or primary Stage IVB carcinoma of the cervix not amenable to curative therapy with either surgery and/or radiation.
* Patients must have biopsy proven squamous cell, adenosquamous, or adenocarcinoma histology.
* Patients do not require measurable disease.
* Patients must have adequate organ function defined by laboratory work.
* Patients must have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Patients must have recovered from any effects attributable to surgery, radiation, or chemoradiotherapy. A minimum of six weeks shall have passed since the last administration of chemoradiotherapy or three weeks for radiation therapy alone.
* Patients must be free of clinically significant infections.
* Patients must be age 19 or greater and have signed informed consent.

Exclusion Criteria:

* Patients who are pregnant or lactating.
* Patients with history of other malignancies (except non-melanoma skin cancer) within the last 5 years are ineligible.
* Patients with non-squamous, adenosquamous, or adenocarcinoma histology.
* Patients with bilateral hydronephrosis that cannot be alleviated by ureteral stents or percutaneous drainage.
* Patients currently receiving any or having received other investigational agents within the last 30 days are ineligible.
* Patients with known hypersensitivity to topotecan or cisplatin.
* Patients with craniospinal metastases.
* Patients with uncontrolled current illness including, but not limited to, ongoing or active infection, unstable angina pectoris, cardiac arrhythmia, serious peripheral neuropathy, or psychiatric illness/social situations that would limit or preclude compliance with study requirements are ineligible.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-07

PRIMARY OUTCOMES:
MTD of topotecan when given weekly with cisplatin

SECONDARY OUTCOMES:
Toxicity profile in patients treated with the combination of topotecan when given weekly with cisplatin
Response rate and time to progression

CONTACTS AND LOCATIONS:
Overall Officials: J. Michael Straughn, Jr., MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States